CLINICAL TRIAL: NCT03663114
Title: A Drug Use Investigation of LENVIMA 4 mg Capsules - A Post-marketing Observational Study on Risk Factors for Hepatic Encephalopathy in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: A Post-marketing Observational Study on Risk Factors for Hepatic Encephalopathy in Participants With Unresectable Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LEN02T; E7080-M081-504 (Other: EISAI)
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; Lenvima; Post-marketing surveillance; LEN02T; Lenvatinib Mesilate
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lenvatinib: Participants receiving lenvatinib capsules 12 milligrams (mg) based on participant's body weight greater than or equal to (>=) 60 kilograms (kg) or 8 mg based on participant's body weight less than (<) 60 kg, orally, once daily dose will be centrally registered and observed prospectively for up to 1 year after the administration of dose.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib capsule
  Other Names: Lenvima; E7080

SUMMARY:
This study is a post-marketing observational study of lenvatinib in participants with unresectable hepatocellular carcinoma. The primary objective of this study is assessment of risk factors for hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with unresectable hepatocellular carcinoma who were administered the lenvatinib mesilate for the first time within the registration period.
* Have provided informed consent.
* Underwent case registration by 14 days after the start of administration of drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants with unresectable hepatocellular carcinoma and administered lenvatinib in Japan will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 713 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Hepatic Encephalopathy Risk Factors | Baseline up to 1 year
  Hepatic encephalopathy risk factors such as constipation, dehydration, infection, gastrointestinal hemorrhage will be assessed.

SECONDARY OUTCOMES:
Number of Participants with Hepatic Encephalopathy | Baseline up to 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Eisai trial site 1, Osaka
  - Eisai trial site 2, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Furuse J, Izumi N, Motomura K, Inaba Y, Katamura Y, Kondo Y, Yabushita K, Matsuoka T, Motoyoshi K, Kudo M. Long-Term Survival of Patients with Unresectable Hepatocellular Carcinoma Treated with Lenvatinib in Real-World Clinical Practice. Cancers (Basel). 2025 Feb 1;17(3):479. doi: 10.3390/cancers17030479. PMID 39941845